CLINICAL TRIAL: NCT00198120
Title: A Randomized Controlled Trial of D-Cycloserine in Autism
Brief Title: Safety and Effectiveness of D-Cycloserine in Children With Autism
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); National Alliance for Research on Schizophrenia and Depression (Other); Indiana University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: K23MH068627 (NIH); K23MH068627 (NIH); 0305-30; DDTR BK-TKND
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2016-04

CONDITIONS: Autistic Disorder
Keywords: Autistic Disorder; cycloserine; pharmacology; glutamatergic agents; communication; social interaction; Double-Blind Method
MeSH Terms: conditions — Autistic Disorder; Communication | interventions — Cycloserine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will receive D-Cycloserine for 8 weeks.
  Interventions: Drug: D-cycloserine
- 2 (Placebo Comparator): Participants will receive placebo for 8 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: D-cycloserine — D-Cycloserine 0.6mg/kg/day in week 1 D-Cycloserine 1.1mg/kg/day in week 2 D-Cycloserine 1.7mg/kg/day in week 3-8 Flexible dosing based on response. Capsule Strength: 10mg, 20mg
  Other Names: Seromycin; Cycloserine
  Arms: 1
Drug: Placebo — Placebo: same dosing schedule and capsule strength
  Arms: 2

SUMMARY:
This study will determine the effectiveness of D-cycloserine in reducing symptoms of autism in autistic children.

DETAILED DESCRIPTION:
This project proposes to study the efficacy and safety of D-cycloserine in children with autism. The central hypothesis of this project is that D-cycloserine will be efficacious in reducing certain symptoms of autism including some aspects of social impairment.

Autism is a severe neuropsychiatric disorder with a prevalence of at least 0.1 %. Despite investigations into the pharmacologic treatment of autism, no drugs have been shown to consistently improve the core symptoms of the disorder, namely social and communication impairment. Pilot data has suggested that D-cycloserine, a drug that affects the N-methyl-D-aspartate (NMDA) subtype of glutamate receptor, has efficacy for the symptom of social withdrawal in autism. In this study, children with autism will be randomly assigned to treatment with either D-cycloserine or placebo for 8 weeks. Both the subjects and investigators will be blind to treatment assignment. Subjects will be rated on a variety of clinical measures to examine the effects of D-cycloserine on social withdrawal and other symptoms of autism. Safety data including side-effects, vital signs, blood tests, and electrocardiograms will be performed at the beginning and end of the study. This study will provide important information about the effects of D-cycloserine for treating core and associated symptoms of autism. It will also greatly expand the knowledge about glutamatergic agents in autism and provide crucial information regarding the pathophysiology and future design of drug studies in autism.

ELIGIBILITY:
Inclusion Criteria:

* Age 3 Years to 12 Years
* Diagnostic Statistical Manual Version -IV (DSM-IV) and Autism Diagnostic Interview - Revised (ADI-R)-confirmed Diagnosis of Autistic Disorder
* Aberrant Behavior Checklist (ABC) Lethargy Subscale Score of 13 or greater

Exclusion Criteria:

* Children with Severe to Profound Mental Retardation
* Weight at Screening Visit <11 kilograms
* Clinical Global Impressions-Severity Score of 7
* Presence of a Neurodevelopmental Disorder with Possible Associations to Autism: Subjects with Fragile X Syndrome, Tuberous Sclerosis, or other neurodevelopmental disorders known to be associated with autism or autistic features will be excluded.
* Presence of a Psychiatric Disorder that would Require a Specific Type of Treatment: Subjects with major depressive disorder, bipolar disorder, or a psychotic disorder will be excluded because treatment for these disorders often requires specific psychotropic agents. Subjects with an active substance use disorder will be excluded because of safety concerns and problems this would cause in assessing efficacy.
* Presence of a Medical Condition that would make Treatment with D-Cycloserine Less Safe: Subjects with significant cardiac, hepatic, or renal disease will be excluded due to concerns about pharmacokinetic alterations or adverse effects. Subjects with epilepsy or a history of seizures will be excluded due to rare reports of seizures with high doses of D-cycloserine. D-cycloserine is an U.S. FDA Pregnancy Category C drug. Because of the unknown effects of D-cycloserine on the developing human fetus, females of childbearing potential will be given a urine pregnancy test and required to use a suitable form of birth control during the study.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2004-02; Primary Completion 2007-09 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Change in Clinical Global Impressions (CGI) Global Improvement | Change from Baseline at 8 Weeks
  All randomized subjects in the Double-Blind Phase will be assessed for change.
Change in Clinical Global Impressions (CGI) Global Improvement | Change from Open-Label Baseline at 8 Weeks
  All placebo non-responders will enter into an open-label phase after the Double-Blind Phase
Change in Lethargy Subscale of the Aberrant Behavior Checklist (ABC) | Change from Baseline at 8 Weeks.
  All randomized subjects in the Double-Blind Phase will be assessed for change.
Change in Lethargy Subscale of the Aberrant Behavior Checklist (ABC) | Change from Open-Label Baseline at 8 Weeks
  All placebo non-responders will enter into an open-label phase after the Double-Blind Phase

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J. McDougle, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Riley Hospital for Children, Christian Sarkine Autism Treatment Center, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Iffland M, Livingstone N, Jorgensen M, Hazell P, Gillies D. Pharmacological intervention for irritability, aggression, and self-injury in autism spectrum disorder (ASD). Cochrane Database Syst Rev. 2023 Oct 9;10(10):CD011769. doi: 10.1002/14651858.CD011769.pub2. PMID 37811711
- [Derived] Aye SZ, Ni H, Sein HH, Mon ST, Zheng Q, Wong YKY. The effectiveness and adverse effects of D-cycloserine compared with placebo on social and communication skills in individuals with autism spectrum disorder. Cochrane Database Syst Rev. 2021 Feb 14;2(2):CD013457. doi: 10.1002/14651858.CD013457.pub2. PMID 33583058